CLINICAL TRIAL: NCT01261767
Title: A Randomised, Double-blind, Placebo-controlled, Single and Multiple Dose, Dose-escalation Trial of Anti-IL-20 (109-0012) 100 mg/Vial in Psoriatic Subjects, Followed by an Expansion Phase
Brief Title: First Human Dose Study of Anti-IL-20 in Psoriasis: A Study of Safety, Tolerability and Early Signals of Biologic and Clinical Effects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Trial discontinued due to apparent lack of response in psoriasis measures. No safety concerns were present
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8226-1848; U1111-1118-2792 (Other: WHO)
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Psoriasis
MeSH Terms: conditions — Inflammation; Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-IL-20 (Experimental)
  Interventions: Drug: anti-IL-20
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: anti-IL-20 — Anti-IL-20 in 100mg/vial for subcutaneous (under the skin) injection
  Arms: Anti-IL-20
Drug: placebo — Placebo for subcutaneous (under the skin) injection
  Arms: Placebo

SUMMARY:
This trial is conducted in the United States of America (USA). The aim of this clinical trial is evaluate the safety and tolerability of anti-IL-20 in patients with psoriasis and to determine the preliminary efficacy in an expansion phase of this trial.

This trial consists of 3 parts: A single dose (SD) dose-escalation phase for 16 weeks, a multiple dose (MD) dose-escalation phase for 22 weeks, and a MD expansion phase for 22 weeks.

Initiation of the MD expansion phase will depend on results from the SD and MD dose-escalation phases and only if an acceptable safety profile is present. Subjects participating in the expansion phase are not allowed to have participated in the previous phases (SD and MD dose-escalation phases) of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with moderate to severe stable chronic plaque psoriasis for at least 6 months, with or without psoriatic arthritis
* Affected body surface area (BSA) greater than or equal to 15%
* Physician's Global Assessment (PGA) score of 3 or more
* Female subjects of non-childbearing potential or postmenopausal for at least 1 year. Male subjects must agree to use effective method of birth control
* Body Mass Index (BMI) less than or equal to 38.0 kg/m2

Exclusion Criteria:

* Concomitant anti-psoriatic treatment
* Infectious disease requiring systemic anti-infectious treatment within the 2 weeks prior to administration of trial drug
* Known history of Human Immunodeficiency Virus (HIV)
* Hepatitis B and/or C (determined by test)
* Live virus or bacteria vaccines within the last month before drug administration
* Known active herpes/herpes zoster/cold sores
* Kidney insufficiency
* Liver insufficiency
* Lymphoproliferative disease
* History or signs of malignancy within the last 5 years

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Observed toxicity using the US National Cancer Institute's common terminology criteria for adverse events (CTCAE) - SD phase | from week 0 until end of trial observation period at week 16
Observed toxicity using the US National Cancer Institute's common terminology criteria for adverse events (CTCAE) - MD and MD expansion phases | from week 0 until end of trial observation period at week 22
Improvement psoriasis area and severity index score by 75% (PASI75) - MD expansion phase | at weeks 1-7, 9-15, 22

SECONDARY OUTCOMES:
Observed toxicity using the US National Cancer Institute's common terminology criteria for adverse events (CTCAE) - MD expansion phase | from week 0 until end of trial observation period at week 22
Improvement psoriasis area and severity index score by 75% (PASI75) - SD and MD phases | SD: at weeks 1, 3, 9, 13 and 16. MD: at weeks 1, 3, 5, 7, 9, 15, 22
Pharmacokinetics (the rate at which the body eliminates the trial drug) - SD and MD phases | SD: Prior to dosing (week 1) and through 24 hours and at each visit (week 1-3, 5, 9, 13 and 16). MD: Prior to dosing and at each dosing visit (week 1, 3, 5, 7)
Pharmacokinetics (the rate at which the body eliminates the trial drug) - MD expansion phase | prior to dosing (week 1) and at each dosing visit (week 2-7)
Pharmacodynamics (the effect of the investigated drug on the body) - SD and MD phases | SD: Prior to dosing (week 1) and through 24 hours and at each visit (week 1-3, 5, 9, 13 and 16). MD: Prior to dosing and at each dosing visit (week 1, 3, 5, 7)
Pharmacodynamics (the effect of the investigated drug on the body) - MD expansion phase | prior to dosing (week 1) and at each dosing visit (week 2-7)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (14):
- United States (14):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Skokie, Illinois
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Baltimore, Maryland
  - Novo Nordisk Investigational Site, Boston, Massachusetts
  - Novo Nordisk Investigational Site, St Louis, Missouri
  - Novo Nordisk Investigational Site, New Brunswick, New Jersey
  - Novo Nordisk Investigational Site, New York, New York
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Portland, Oregon
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, Norfolk, Virginia

REFERENCES:
- [Result] Lundblad MS, Overgaard RV, Gothberg M, Fjording MS, Watson E. Clinical pharmacokinetics of the anti-interleukin-20 monoclonal antibody NNC0109-0012 in healthy volunteers and patients with psoriasis or rheumatoid arthritis. Adv Ther. 2015 Mar;32(3):228-38. doi: 10.1007/s12325-015-0191-7. Epub 2015 Mar 7. PMID 25749867
- [Derived] Gottlieb AB, Krueger JG, Sandberg Lundblad M, Gothberg M, Skolnick BE. First-In-Human, Phase 1, Randomized, Dose-Escalation Trial with Recombinant Anti-IL-20 Monoclonal Antibody in Patients with Psoriasis. PLoS One. 2015 Aug 7;10(8):e0134703. doi: 10.1371/journal.pone.0134703. eCollection 2015. PMID 26252485
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com